CLINICAL TRIAL: NCT01649895
Title: Internet-based Cognitive Behavior Therapy in Combination With D-Cycloserine for Obsessive Compulsive Disorder: A Double Blinded Randomized Controlled Trial
Brief Title: D-Cycloserine as an Adjunct to Internet-CBT for OCD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Christian Rück (Other)
Collaborators: The Swedish Research Council (Other Government); Königska (Unknown); Region Stockholm (Other Government)
Responsible Party: Sponsor-Investigator, Christian Rück, MD, PhD, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-002819-28
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Obsessive-compulsive Disorder
Keywords: Obsessive-compulsive disorder; internet; cognitive-behaviour therapy; D-Cycloserine
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cycloserine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-Cycloserine (Experimental): D-Cycloserine, 5 pills (50mg), once per week in 5 weeks.
  Interventions: Drug: D-Cycloserine
- Placebo (Placebo Comparator): Placebo: 5 pills for 5 weeks, once per week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-Cycloserine — Predicted to enhance the effects of exposure in internet-based cognitive-behaviour therapy
  Other Names: DCS; C3H6N2O2; Cycloserine
  Arms: D-Cycloserine
Drug: Placebo — Placebo pills as adjunct to internet-based cognitive-behaviour therapy
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine if D-Cycloserine is an effective adjunct to internet-based cognitive behaviour therapy for patients with obsessive-compulsive disorder.

DETAILED DESCRIPTION:
Trial Objectives:

Primary aim is to investigate whether D-Cycloserine gives incremental effects to ICBT in terms of reduced OCD symptoms. Secondary aims are to a) replicate previous findings in that DCS fastens the effects of CBT, b) correlate the fastened effect to overall treatment adherence and c) investigate gene variation and therapeutic factors as predictors of symptom severity, symptom type and treatment response.

Trial Design: Double blinded randomized controlled trial

Dose/Duration: 5 capsules of 50 mg D-Cycloserine or placebo. 1 pcs per week for 5 weeks. All participants also receive Internet-based cognitive behavior therapy for 12 weeks.

Primary Endpoint: Change from W0-W13 and 3-months follow-up.

Efficacy Parameters: Y-BOCS clinician rated.

Safety Parameters: Adverse Events assessed weekly via the internet and also at post-treatment and at 3-months follow-up using face-to-face clinician assessments.

Description of Trial Subjects: Fulfilling diagnostic criteria of OCD not associated with hoarding.

Number of Subjects: 128

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Male or female
* ≥ 18 years
* Currently living in Stockholm, Uppland, Örebro, Södermanland, Gästrikland, Västmanland and Östergötland county in Sweden.
* Primary diagnosis of OCD according to the DSM-IV-TR.
* Signed informed consent
* Have regular access to a computer with internet access and skills to use the web
* Have received information about the need of using contraception

Exclusion Criteria:

* Pregnancy or breast feeding
* Patients unlikely to cooperate fully in the study
* Patients not able to read or understand the basics of the ICBT self-help material
* Psychotropic medication changes within two months prior to treatment
* Completed CBT for OCD within last 12 months
* Y-BOCS [21] < 16 at Psychiatrist visit (6.2.3)pi
* OCD symptoms primarily associated with hoarding.
* Other primary axis I diagnosis according to the Mini-International Neuropsychiatric Interview (MINI) [34]
* Ongoing substance dependence
* Lifetime bipolar disorder or psychosis
* Suicidal ideation
* Axis II diagnosis that could jeopardize treatment participation
* Serious physical illness that will be an obstacle in ICBT and DCS
* Other ongoing psychological treatments that could affect OCD symptoms
* Epilepsia
* Renal impairment
* Hypersensitivity to D-Cycloserine
* Porphyria
* Chronic Alcoholism

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (Y-BOCS) (clinician rated) | W0,W6,W13. Mid assessments immediately before and after DCS treatment. Long term follow-up at 3-, 12- and 24 months after treatment has ended
  Change from Baseline in OCD severity after 12 weeks and at 3-, 12- and 24 months after treatment has ended.

SECONDARY OUTCOMES:
Obsessive Compulsive Scale - Revised (OCI-R) | W0, W13, Long term follow-up at 3-, 12- and 24 months after treatment has ended
  Change from Baseline in OCD severity after 12 weeks and at 3-, 12- and 24 months after treatment has ended.
Yale Brown Obsessive Compulsive Scale (Y-BOCS)(self-rated) | W0, W1,W2,W3,W4,W5,W6,W7,W8,W9,W10,W11,W12, Long term follow-up at 3-, 12- and 24 months after treatment has ended
  Weekly change from Baseline in OCD severity during 12 weeks of treatment and at 3-, 12- and 24 months after treatment has ended.
Montgomery Asberg Depression Rating Scale Self-rating (MADRS-S) | W0, W13, Long term follow-up at 3-, 12- and 24 months after treatment has ended
  Change from Baseline in depression after 12 weeks and at 3-, 12- and 24 months after treatment has ended.
Euroqol | W0, W13, Long term follow-up at 3-, 12- and 24 months after treatment has ended
  Change from Baseline in quality of life after 12 weeks and at 3-, 12- and 24 months after treatment has ended.
Trimbos and institute of medical technology assessment cost questionnaire for psychiatry (TIC-P) | W0, W13, Long term follow-up at 3-, 12- and 24 months after treatment has ended
  Change from Baseline in societal costs after 12 weeks and at 3-, 12- and 24 months after treatment has ended.
Global assessment of functioning (GAF) | W0, W13, Long term follow-up at 3-, 12- and 24 months after treatment has ended
  Change from Baseline global functioning after 12 weeks and at 3-, 12- and 24 months after treatment has ended.
Clinical global impression (CGI) | W0, W13, Long term follow-up at 3-, 12- and 24 months after treatment has ended
  Change from Baseline in Clinical global impression after 12 weeks and at 3-, 12- and 24 months after treatment has ended.
Adverse events | W0, W1,W2,W3,W4,W5,W6,W7,W8,W9,W10,W11,W12,W13 Long term follow-up at 3-, 12- and 24 months after treatment has ended
  Weekly adverse events reporting during 12 weeks of treatment and at 3-, 12- and 24 months after treatment has ended.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rück, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- M46 Huddinge sjukhus, Internetpsykiatrienheten/mottagningen för tvångssyndrom, Stockholm, Sweden

REFERENCES:
- [Result] Andersson E, Hedman E, Enander J, Radu Djurfeldt D, Ljotsson B, Cervenka S, Isung J, Svanborg C, Mataix-Cols D, Kaldo V, Andersson G, Lindefors N, Ruck C. D-Cycloserine vs Placebo as Adjunct to Cognitive Behavioral Therapy for Obsessive-Compulsive Disorder and Interaction With Antidepressants: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Jul;72(7):659-67. doi: 10.1001/jamapsychiatry.2015.0546. PMID 25970252